CLINICAL TRIAL: NCT06974266
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Preliminary Efficacy of Akkermansia Muciniphila AKM Lab-01 in Subjects With Hypercholesterlemia
Brief Title: An Efficacy and Safety Study of Akkermansia Muciniphila AKM Lab-01 in Hypercholesterolaemia
Acronym: AKM Lab-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moon (Guangzhou) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MN-AKM-101
Record Dates: First submitted 2025-04-14; First posted 2025-05-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Subjects receive AKM Lab-01 Enteric-coated Capsule
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Subjects receive placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Subjects receive AKM Lab-01 Enteric-coated once daily by oral, 34B TFU/day , within half an hour after breakfast for 3 months.
  Arms: Probiotic
Dietary Supplement: Placebo — Subjects receive placebo once daily by oral, one capsule/day, within half an hour after breakfast for 3 months.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the safety and efficacy of AKM Lab-01 in subjects with hypercholesterolemia. This study will be conducted as a randomized, double-blind, placebo-controlled trial, eligible hypercholesterolemic participants were administered daily oral doses of either AKM Lab-01 or a placebo. Baseline clinical parameters, blood samples, and stool specimens were collected before and after the intervention for comparative analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-60 years (inclusive), regardless of gender;
2. Patients diagnosed with hypercholesterolemia (5.2 mmol/L ≤ TC <6.2 mmol/L, or 3.4 mmol/L ≤ LDL-C <5.0 mmol/L), with or without hypertriglyceridemia (1.7 mmol/L ≤ TG <4.5 mmol/L) or mixed hyperlipidemia (defined as: 1.7 mmol/L ≤ TG <4.5 mmol/L and 5.2 mmol/L ≤ TC <6.2 mmol/L; or 1.7 mmol/L ≤ TG <4.5 mmol/L and 3.4 mmol/L ≤ LDL-C <5.0 mmol/L; or 1.7 mmol/L ≤ TG <4.5 mmol/L, 5.2 mmol/L ≤ TC <6.2 mmol/L and 3.4 mmol/L ≤ LDL-C <5.0 mmol/L);
3. Accompanied by overweight/obesity (24.0 ≤ BMI ≤40.0 kg/m²);
4. Have not taken any metabolic control medications (for lipid, weight, or blood glucose) within the past month;
5. Have controlled of blood lipids solely through lifestyle interventions (diet and exercise) for at least 1 month prior to the screening period;
6. People must possess communication and cognitive abilities to adhere to long-term medication, and fully understand the nature, significance, potential benefits, inconveniences, and risks of the study before participation;
7. Fertile patients (male or female) must agree to use at least one medically approved contraceptive method (e.g., intrauterine device [IUD], oral contraceptives, or condoms) during the trial. Female with childbearing potential must have a negative blood pregnancy test during screening and must not be lactating;
8. Voluntary enrollment with signed informed consent, and commitment to comply with the trial treatment regimen and visit schedule

Exclusion Criteria:

1. Have taken any metabolic control medications (e.g., lipid-lowering, blood glucose-regulating, or weight-loss drugs) within the past month or are currently taking such medications.
2. Patients with secondary hyperlipidemia caused by conditions such as nephrotic syndrome, liver diseases, hypothyroidism, renal failure, etc..
3. Have severe comorbidities requiring immediate treatment, including uncontrolled diabetes, hypertriglyceridemia, cerebrovascular diseases, etc., as determined by the investigator.
4. Have severe primary diseases (e.g., hepatic, renal, or hematopoietic system disorders) or psychiatric conditions.
5. Patients with a family history of genetically inherited metabolic disorders.
6. Currently taking liver-affecting medications.
7. Have a history of bariatric surgery.
8. People with acute or chronic progressive/unstable diseases deemed unsuitable for enrollment by the investigator.
9. Hepatic or renal dysfunction: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5×upper limit of normal (ULN); Total bilirubin >1.5×ULN; Serum creatinine (Cr) >1.5×ULN.
10. Serum amylase ≥1.5×ULN or other clinically significant laboratory abnormalities per investigator judgment.
11. Patients with acute diabetic complications (e.g., diabetic ketoacidosis, hyperosmolar hyperglycemic state) within the past 3 months.
12. Have a history of gastrointestinal surgery within the past year.
13. People with allergic constitution or hypersensitivity to the investigational product.
14. Have used antibiotics, probiotics, or prebiotics within 3 months prior to recruitment.
15. Excessive alcohol consumption in the past decade (>30 g/day for males; >20 g/day for females).
16. Pregnant or breastfeeding subjects.
17. Excluded for other reasons as determined by the investigator.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in TC and LDL-C | Baseline, Day30，Day90
  The changes in serum TC and LDL-C of participants from baseline
AE and SAE | Up to 4months
  During the trial, all subjects are observed and recorded for any adverse events (AEs) that occur during the study period, the incidence, type and severity of serious adverse events (SAEs), including clinical symptoms and abnormalities in vital signs, and abnormalities in lab tests, with determination of the correlation between them and the investigational drug.

SECONDARY OUTCOMES:
Changes in Blood Lipids | Baseline, Day30, Day90
  Changes of participants from baseline in HDL-C and Triglyceride
Changes in FBG | Baseline, Day30, Day90
  Changes of participants from baseline in Fasting blood glucose (FBG)
Changes in Blood Pressure | Baseline, Day30, Day90
  Changes of participants from baseline in blood pressure
Changes in Uric Acid | Baseline, Day30, Day90
  Changes of participants from baseline in Uric Acid
Changes in Weight | Baseline, Day30, Day90
  Changes of participants from baseline in weight
Changes in HbA1c | Baseline, Day30, Day90
  Changes of participants from baseline in HbA1c
Changes in Waist Circumference and Hip Circumference | Baseline, Day30, Day90
  Changes of participants from baseline in waist circumference and hip circumference
Changes in Body Fat Percentage | Baseline, Day30, Day90
  Changes of participants from baseline in body fat percentage

CONTACTS AND LOCATIONS:
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided